CLINICAL TRIAL: NCT05641324
Title: A Phase 1 Study of ANV419 as Monotherapy, and ANV419 in Combination With Daratumumab or With Lenalidomide Plus Low-Dose Dexamethasone, in Patients With Relapsed or Refractory Multiple Myeloma (OMNIA-2)
Brief Title: A Study of ANV419 Alone or in Combination With Approved Treatments in Patients With Multiple Myeloma (OMNIA-2)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was ended due to a lack of recruitment
Sponsor: Anaveon AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ANV419-102
Record Dates: First submitted 2022-11-29; First posted 2022-12-07 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Multiple Myeloma; Relapsed Cancer; Refractory Multiple Myeloma; Adult Disease; Hematologic Diseases
Keywords: IL-2; ANV419; Cancer; Multiple Myeloma; OMNIA
MeSH Terms: conditions — Multiple Myeloma; Recurrence; Disease; Hematologic Diseases; Neoplasms | interventions — Lenalidomide; Dexamethasone; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ANV419 single agent, dose 1, Q2W (Experimental)
  Interventions: Drug: ANV419
- ANV419 single agent, dose 2, Q2W (Experimental)
  Interventions: Drug: ANV419
- ANV419 Q2W + Lenalidomide plus low-dose dexamethasone (Experimental)
  Interventions: Drug: ANV419; Drug: Lenalidomide with low-dose dexamethasone
- ANV419 Q2W + Daratumumab (Experimental)
  Interventions: Drug: ANV419; Drug: Daratumumab

INTERVENTIONS:
Drug: ANV419 — ANV419 administered by intravenous (IV) infusion
Drug: Lenalidomide with low-dose dexamethasone — Lenalidomide and dexamethasone administered orally
  Arms: ANV419 Q2W + Lenalidomide plus low-dose dexamethasone
Drug: Daratumumab — Daratumumab administered by subcutaneous injection
  Arms: ANV419 Q2W + Daratumumab

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of ANV419 monotherapy followed by ANV419 in combination with lenalidomide plus low-dose dexamethasone or ANV419 in combination with daratumumab.

DETAILED DESCRIPTION:
The purpose of this multi-site, open-label, Phase 1 adaptive design study is to evaluate the safety, tolerability and preliminary efficacy of ANV419 as a monotherapy followed by ANV419 in combination with lenalidomide plus low-dose dexamethasone or ANV419 in combination with daratumumab in patients aged 18 years or older with with relapsed or refractory Multiple Myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Must provide written informed consent for the study;
* Must be able to comply with the Protocol as judged by the Investigator;
* Are ≥18 years of age on the day of signing informed consent
* Have been diagnosed with symptomatic MM per CRAB (calcium elevation, renal dysfunction, anemia, bone disease) criteria;
* Have had evidence of a response (defined as partial response [PR] or better according to IMWG response criteria [Appendix C]) during previous treatment;
* Have undergone treatment with ASCT or have progressed from at least 2 other prior treatment lines (including an immunomodulatory imide drug and/or daratumumab);
* Have relapsed on, or been refractory or intolerant to, the last treatment line, and have measurable disease evaluated by monoclonal proteins (M-proteins) and/or free light chains according to IMWG response criteria (Appendix C). Non-secretory MM must have measurable, active lesions by positron emission tomography;
* Have a performance status of 0 to 2 on the ECOG Performance Status;
* Have adequate organ functions;
* Willing to undergo bone marrow biopsies if determined clinically feasible based on the Investigator's assessment;
* Are eligible for treatment with daratumumab;
* Are eligible for treatment or re-treatment with lenalidomide (as per the European Medicines Agency labeling criteria);
* Are eligible for prophylaxis for thromboembolism per IMWG response criteria;
* Female patients of childbearing potential must have a negative serum pregnancy test at screening and a negative (urine or serum) pregnancy test within 72 hours prior to receiving the first dose of study drug. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required and must be negative for the patient to be eligible;
* Female patients who are not postmenopausal, and who have not undergone surgical sterilization, must agree to use highly effective methods of contraception during the treatment period and for 6 months after the last dose of study drug. They must also agree not to donate eggs (ova, oocytes) during the same timeframe; and
* Male patients with partners of childbearing potential must agree to use highly effective methods of contraception and barrier contraception (condom) during the treatment period and for 6 months after the last dose of study drug. They must also agree not to donate sperm during the same timeframe.

Exclusion Criteria:

* Have received an investigational agent (including investigational device) <4 weeks or 5 half-lives prior to study Cycle 1 Day 1, whichever is longer;
* Have hypersensitivity to any components of ANV419 (IL-2, anti-IL-2 mAb) or its formulation (L-histidine, L-histidine HCl, sucrose, polysorbate 80, water; see Appendix D);
* Have hypersensitivity to lenalidomide, dexamethasone, daratumumab, or any of their excipients;
* Have received daratumumab <3 months prior to the signing of informed consent;
* Have received any drugs that may be active for MM <3 weeks prior to the signing of informed consent;
* Have received high-dose corticosteroids (≥1 mg/kg) ≤3 weeks prior to the signing of informed consent;
* Have received radiotherapy ≤1 month prior to the signing of informed consent;
* Have had an autologous hematopoietic cell transplant (HCT) within the last 6 months;
* Have had a previous allogeneic HCT;
* Have had major surgery <4 weeks prior to the signing of informed consent or anticipate the need for major surgery during treatment; Note: Major surgery is defined as any surgery requiring entrance into a body cavity (eg, chest, abdomen, or brain), organ removal, normal anatomy alteration, or joint replacement. Minor surgery is defined as any surgery in which skin, mucosa, or connective tissue sections are altered (eg, biopsy, cataract, endoscopic procedures, etc).
* Have clinical signs of meningeal involvement of MM;
* Have a history of a past or current malignancy prior to screening, except for:

  1. Cervical carcinoma of Stage 1B or less;
  2. Non-invasive basal cell or squamous cell skin carcinoma requiring treatment; or
  3. Current or past malignancy with a complete response for <3 years at screening.
* Have plasma cell leukemia defined as a plasma cell count >2000/mm3;
* Have known amyloidosis;
* Have sensory and/or motor neuropathy ≥Grade 3 per NCI CTCAE version 5.0 at screening;
* Have active (measurable) and/or uncontrolled (unresponsive to current therapy) infectious disease (bacterial, fungal, viral, or protozoic);
* Have evidence of uncontrolled (unresponsive to current therapy), concomitant disease including, but not limited to, uncontrolled diabetes mellitus (pre-existing diabetes mellitus type 1 is acceptable), chronic obstructive pulmonary diseases Grade 3 (per NCI CTCAE version 5.0) or higher, asthma, bronchospasm, obstructive pulmonary disease, hematological diseases except MM, renal impairment (except when related to MM), hyperthyroidism due to thyroiditis, known autoimmune disease, or disease with ongoing fibrosis;
* Have clinically significant (defined as a disease that requires intervention) cardiovascular disease including, but not limited to, acute myocardial infarction and/or transient ischemic attack <6 months prior to screening, unstable angina, congestive heart failure (New York Heart Association Class II or higher), or arrhythmia requiring therapy;
* Have an average QTcF interval >480 msec at screening;
* Have active, untreated, immune-related endocrinopathy untreatable with hormone replacement or prior immune-related toxicities (eg, colitis, neuropathy) >Grade 3 (per NCI CTCAE version 5.0) after treatment with immunostimulatory drugs that have not been resolved;
* Have evidence of severe hepatic impairment (equivalent to Child-Pugh Class C [for liver cirrhosis] or a MELD [Model for End-Stage Liver Disease] score of 10 or higher for hepatic impairment not limited to cirrhosis]);
* Have a history or current evidence of any condition, therapy, or laboratory abnormality that might significantly confound the results of the study, interfere with the patient's participation for the full duration of the study, or it is not in the best interest of the patient to participate in the study, in the opinion of the treating Investigator;
* Have a known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the study;
* Are pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, from screening through 6 months after the last dose of study drug;
* Are known to be human immunodeficiency virus (HIV) positive (or tests positive for HIV 1 or 2 at screening), unless the following criteria are met:

  1. CD4+ lymphocyte count >350 µL;
  2. Had no history of AIDS (acquired immunodeficiency syndrome)-defining opportunistic infections within the past 12 months;
  3. Have been on established anti-retroviral therapy for at least 4 weeks; and
  4. Have an HIV viral load of <400 copies/mL prior to study Day 1. Note: Patients on strong cytochrome P450 (CYP)3A4 inhibitors or strong CYP3A4 inducers must be switched to an alternate effective anti-retroviral therapy regimen prior to study treatment or are excluded if regimen prior to study Day 1 cannot be altered.
* Have uncontrolled hepatitis B infection or hepatitis C infection; Note: Patients with hepatitis B (positive hepatitis B surface antigen) who have controlled infection (serum hepatitis B virus DNA by PCR that is below the limit of detection and receiving anti-viral therapy for hepatitis B) are permitted. Patients with controlled infections must undergo periodic monitoring of hepatitis B virus DNA. Note: Patients with hepatitis C (positive hepatitis C virus antibody) who have controlled infection (undetectable hepatitis C virus RNA by PCR either spontaneously or in response to a successful prior course of anti-hepatitis C virus therapy) are permitted.
* Have received a live vaccine within 30 days of study Day 1. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (eg, Flu-Mist®) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) with ANV419 monotherapy | Day 1 up to 12 months
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) with ANV419 in combination with lenalidomide plus low-dose dexamethasone | Day 1 up to 12 months
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) with ANV419 in combination with daratumumab | Day 1 up to 12 months

SECONDARY OUTCOMES:
Serum concentration of ANV419 in blood | Day 1 up to 12 months
Impact of ANV419 on the expression of markers of PBMC lineage in blood | Day 1 up to 12 months
Levels of specific anti-ANV419 antibodies in blood | Day 1 up to 12 months
Objective Response Rate (ORR) as defined by IMWG response criteria, with ANV419 monotherapy | Day 1 up to 12 months
Objective Response Rate (ORR) as defined by IMWG response criteria, with ANV419 in combination with lenalidomide plus low-dose dexamethasone | Day 1 up to 12 months
Objective Response Rate (ORR) as defined by IMWG response criteria, with ANV419 in combination with daratumumab | Day 1 up to 12 months
Quality of life assessed with European Quality of Life Five Dimensions Questionnaire (EQ-5D-5L) | Day 1 up to 12 months
Quality of life assessed with European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Day 1 up to 12 months
Progression-free survival (PFS) according to IMWG response criteria | Day 1 up to 12 months
Duration of Response (DOR) according to IMWG response criteria | Day 1 up to 12 months
Clinical Benefit Rate (CBR) according to IMWG response criteria | Day 1 up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Gasal, MD, Study Director — Anaveon AG
Locations (11):
- Vejle Hospital, Vejle, Denmark
- France (3):
  - Institut Paoli-Calmettes, Marseille
  - CHU de Nantes - Hôtel-Dieu, Nantes
  - Institut de cancérologie Strasbourg Europe (ICANS), Strasbourg
- Universitätsklinikum Jena, Jena, Germany
- Spain (4):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitario La Princesa, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Clinico Universitario de Salamanca, Salamanca
- Switzerland (2):
  - Inselspital, Universitätsspital Bern, Bern
  - Kantonsspital St. Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No